CLINICAL TRIAL: NCT01920646
Title: The Effect of African Leafy Vegetables on Nutritional Status (Including Iron, Zinc and Vitamin A Status) of School Children Residing in Semi-rural Farm Community in the North West Province of South Africa
Brief Title: Effect of African Leafy Vegetables on Nutritional Status of South African School Children.
Acronym: ALV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North-West University, South Africa (Other)
Collaborators: Medical Research Council, South Africa (Other); Agricultural Research Council of South Africa (Unknown); Sight and Life (Unknown); Program to Support Pro-poor Policy Development (PSPPD) (Unknown); National Research Foundation of South Africa (Other)
Responsible Party: Principal Investigator, Marinka van der Hoeven, Mrs Marinka van der Hoeven, North-West University, South Africa
Allocation: Randomized
Other Study IDs: ALV study
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Iron Status; Vitamin A Status; Zinc Status; Malnutrition
MeSH Terms: conditions — Malnutrition

ARMS (2):
- ALV (Experimental): 300 gram cooked African leafy vegetables and school meal starch as daily school meal (5 days/weeks) for 3 months.
  Selected African leafy vegetables:Amaranthus cruentus (amaranth), Vigna unguiculata (cowpea), Cleome gynandra (spiderplant), and Cucurbita maxima (pumpkin).
  Interventions: Other: ALV
- Control (No Intervention): normal school meal as daily meal (5 days/weeks) for 3 months

INTERVENTIONS:
Other: ALV — Random allocation of children of two rural farm schools per grade to receive either 300 gram cooked ALVs and school meal starch or the normal school meal as daily meal (5 days/weeks) for 3 months.
  Arms: ALV

SUMMARY:
The combination of poverty-related infectious and lifestyle-related non-communicable diseases, both driven by malnutrition, causes a high burden for South Africa. Healthy and nutritious diets for populations depend on availability and accessibility of a variety of plant and animal foods, within a context that promotes and supports healthy behaviour. Food based strategies, such as supplementation, food fortification, and diversification of crops, are used to achieve optimal dietary requirements to combat malnutrition, including micronutrient deficiencies. A more sustainable food based strategy is the (promotion of) use of indigenous and traditional foods, such as African Leafy Vegetables (ALVs). Unfortunately, several studies from all over Africa have shown that there is a shift from traditional diets as result of the preparing techniques and the absence of women in homes. Furthermore, indigenous and traditional foods are considered as "poor people's food".

Against this background, a joint project between South Africa, Kenya and Benin is designed to fill the gaps in knowledge in these countries regarding the availability, acceptability and consumption and evidenced based benefits of foods from local biodiversity. The main aim of the study in South Africa is to provide empirical evidence of how the role of biodiversity can be translated into improved health status in contemporary poor rural and urban communities in the North West Province of South Africa. In order to achieve this it is important to gain knowledge on the possibility of using ALVs as a strategy to alleviate micronutrient deficiencies. Therefore an intervention study to determine the effect of selected ALV on the nutritional status (including zinc, iron, and vitamin A status) of school children (grade R-4) residing in contemporary poor rural community in the North West Province, South Africa has been designed.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy and had no signs and symptoms of acute illness at the time of baseline blood collection
* attending grade R - 4 of one of the selected schools

Exclusion Criteria:

* Children with a haemoglobin concentration <8 g/dL were excluded from the study and referred for medical treatment.
* Children who received micronutrient supplements were also excluded from the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in nutritional status of school children (nutritional status measured by: blood haemoglobin, serum ferritin, serum zinc and serum retinol) | three months

SECONDARY OUTCOMES:
Change in nutritional status of school children (nutritional status measured by: height-for-age z-score, weight-for-age z-score and BMI-for-age z-score) | three months

CONTACTS AND LOCATIONS:
Overall Officials: Marius Smuts, PhD, Study Director — North-West University; Annamarie Kruger, PhD, Study Director — North-West University; Marinka van der Hoeven, MSc, Principal Investigator — North-West University
Locations (1):
- Sizamela Intermediate School and Buffelsvlei Intermediate School, Rysmierbult, North West, South Africa